CLINICAL TRIAL: NCT07245459
Title: The Effect of a Cardiac Rehabilitation Program Including Moderate-Intensity Continuous Exercise Training and High-Intensity Interval Exercise Training on Sarcopenia and Myokines in Patients With Heart Failure
Brief Title: Cardiac Rehabilitation in Heart Failure and Sarcopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Collaborators: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Ebru Alemdaroğlu, Ankara Bilkent City Hospital, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E2-24-7194
Record Dates: First submitted 2025-11-13; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure
Keywords: heart failure; cardiac rehabilitation; sarcopenia; Myokines
MeSH Terms: conditions — Heart Failure; Sarcopenia | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patients will be blinded to group allocation, and the exercise group will be determined through randomization, after which the appropriate program will be administered accordingly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIT (high intensity interval training) (Experimental): For the HIIT group, the first week consists of three sessions including a 5-minute warm-up at 30% of VO₂max, 20 minutes of exercise at 60% of VO₂max, and a 5-minute cool-down at 30% of VO₂max. Starting from the second week, interval training will be implemented as follows: 5 sessions of 20 minutes with intervals alternating between 65-80% of VO₂max for 60 seconds and 50% of VO₂max for 120 seconds; 5 sessions of 20 minutes alternating 65-80% of VO₂max for 120 seconds and 50% of VO₂max for 120 seconds; and 5 sessions of 20 minutes alternating 65-80% of VO₂max for 240 seconds and 50% of VO₂max for 180 seconds.
  Interventions: Other: HIIT (high intensity interval training)
- MCT (moderate intensity continuous training) (Experimental): For the MCT group, the program will be included a 5-minute warm-up at 30% of VO₂max, followed by 20 minutes of continuous exercise at 60% of VO₂max, and a 5-minute cool-down at 30% of VO₂max.
  Interventions: Other: MCT (moderate intensity continuous training)

INTERVENTIONS:
Other: HIIT (high intensity interval training) — For the HIIT group, the first week consists of three sessions including a 5-minute warm-up at 30% of VO₂max, 20 minutes of exercise at 60% of VO₂max, and a 5-minute cool-down at 30% of VO₂max. Starting from the second week, interval training will be implemented as follows: 5 sessions of 20 minutes with intervals alternating between 65-80% of VO₂max for 60 seconds and 50% of VO₂max for 120 seconds; 5 sessions of 20 minutes alternating 65-80% of VO₂max for 120 seconds and 50% of VO₂max for 120 seconds; and 5 sessions of 20 minutes alternating 65-80% of VO₂max for 240 seconds and 50% of VO₂max for 180 seconds
  Arms: HIIT (high intensity interval training)
Other: MCT (moderate intensity continuous training) — For the MCT group, the program will be included a 5-minute warm-up at 30% of VO₂max, followed by 20 minutes of continuous exercise at 60% of VO₂max, and a 5-minute cool-down at 30% of VO₂max.
  Arms: MCT (moderate intensity continuous training)

SUMMARY:
In this study, it is aimed to investigate the effects of a cardiac rehabilitation program consisting of two different aerobic exercise modalities on aerobic capacity, symptoms, quality of life, and sarcopenia in patients with heart failure who present with one or more symptoms such as dyspnea, difficulty walking, muscle weakness, or limitations in activities of daily living and who are in need of cardiac rehabilitation.

DETAILED DESCRIPTION:
Patients who were followed up in the Heart Failure Clinic, aged 18-75, had stable clinical symptoms, and were referred to Cardiopulmonary Rehabilitation Unit for the cardiac rehabilitation program and met the inclusion criteria will be included in our study.

Prior to initiating the program, participants will be prescribed an individualized exercise regimen determined to be both effective and safe, based on their exercise capacity assessed through the CPET-derived optimal exercise prescription. For the MCT group, the program includes a 5-minute warm-up at 30% of VO₂max, followed by 20 minutes of continuous exercise at 60% of VO₂max, and a 5-minute cool-down at 30% of VO₂max.

For the HIIT group, the first week consists of three sessions including a 5-minute warm-up at 30% of VO₂max, 20 minutes of exercise at 60% of VO₂max, and a 5-minute cool-down at 30% of VO₂max. Starting from the second week, interval training will be implemented as follows: 5 sessions of 20 minutes with intervals alternating between 65-80% of VO₂max for 60 seconds and 50% of VO₂max for 120 seconds; 5 sessions of 20 minutes alternating 65-80% of VO₂max for 120 seconds and 50% of VO₂max for 120 seconds; and 5 sessions of 20 minutes alternating 65-80% of VO₂max for 240 seconds and 50% of VO₂max for 180 seconds.

Both groups will be completed a total of 18 sessions over 6 weeks, with training occurring three times per week. Resistance training exercises will be incorporated into the programs in both groups after the second week. Load increments of 5 watts will be applied based on patient tolerance.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18-75 years heart failure (HF) NYHA class II-III left ventricular ejection fraction (LVEF) <0.40, BMI between 18-30 kg/m² standard medications at stable doses for at least two weeks prior to enrollment

-

Exclusion Criteria:

a history of cardiac implant device placement within the previous 6 weeks a planned cardiac device implantation heart transplantation within the next 12 months acute coronary syndrome within the prior 6 weeks severe valvular or congenital heart disease severe hypertrophic obstructive cardiomyopathy acute myocarditis or pericarditis intracardiac thrombus primary pulmonary hypertension peripartum cardiomyopathy uncontrolled hypertension (systolic blood pressure >200 mmHg and/or diastolic blood pressure >110 mmHg) severe arrhythmias.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
VO2 max | Day 1 and 6th week
  The maximal oxygen uptake (VO2max) in Cardiopulmonary exercise test (CPET)

SECONDARY OUTCOMES:
Myostatin | Day 1 and 6th week
BDNF | Day 1 and 6th week

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Q, Zhang L, Zhang Z, Wang Y, Zuo C, Bo S. A Shorter-Bout of HIIT Is More Effective to Promote Serum BDNF and VEGF-A Levels and Improve Cognitive Function in Healthy Young Men. Front Physiol. 2022 Jun 29;13:898603. doi: 10.3389/fphys.2022.898603. eCollection 2022. PMID 35846013
- [Background] Donelli da Silveira A, Beust de Lima J, da Silva Piardi D, Dos Santos Macedo D, Zanini M, Nery R, Laukkanen JA, Stein R. High-intensity interval training is effective and superior to moderate continuous training in patients with heart failure with preserved ejection fraction: A randomized clinical trial. Eur J Prev Cardiol. 2020 Nov;27(16):1733-1743. doi: 10.1177/2047487319901206. Epub 2020 Jan 21. PMID 31964186
- [Background] Springer J, Springer JI, Anker SD. Muscle wasting and sarcopenia in heart failure and beyond: update 2017. ESC Heart Fail. 2017 Nov;4(4):492-498. doi: 10.1002/ehf2.12237. PMID 29154428